CLINICAL TRIAL: NCT06827223
Title: Comparative Evaluation of the Effect of Computer-controlled Starpen Automatic Injection Device Versus Traditional Syringe on Pain Perception During Nerve Block Anesthesia and Extraction of Mandibular Primary Molars: a Randomized Controlled Trial
Brief Title: Effect of Starpen CCLAD in Injection and Extraction
Acronym: Starpen CCLAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Mostafa Abohashim Masoud Soliman, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Starpen CCLAD in injection
Record Dates: First submitted 2025-01-25; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Pain Assessment
Keywords: Starpen CCLADS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): nerve block anesthesia and extraction of mandibular primary molars using a Traditional Syringe
  Interventions: Device: Traditional Syringe
- intervention group (Experimental): nerve block anesthesia and extraction of mandibular primary molars using Computer-controlled Starpen Automatic Injection Device
  Interventions: Device: computer-controlled Starpen Automatic Injection Device

INTERVENTIONS:
Device: computer-controlled Starpen Automatic Injection Device — using computer-controlled Starpen Automatic Injection Device during inferior alveolar nerve block anesthesia and extraction of mandibular primary molars
  Arms: intervention group
Device: Traditional Syringe — nerve block anesthesia and extraction of mandibular primary molars using Traditional Syringe
  Arms: control group

SUMMARY:
The present study aims to evaluate the effect of computer-controlled Starpen automatic injection device versus the traditional syringe on pain perception during Injection of nerve block anesthesia and extraction of mandibular primary molars.

DETAILED DESCRIPTION:
Pain is "An unpleasant sensory and emotional experience connected to actual or potential tissue damage or described in terms of such damage". According to the American Academy of Pediatric Dentistry, a patient may experience serious physical and psychological complications from improper pain management.

Anxiety, a fear of dental procedures, is often linked to unpleasant stimuli such as needle phobia, high vibration, noises, pain, and the smell of materials or medications. Patients who experience anxiety often exhibit complex behavior before or during dental procedures, causing additional discomfort.

In most dental procedures, Local anesthetic (LA) is crucial to alleviate pain during dental procedures enabling the dentist to complete the process. Even though LA is used to reduce pain during the procedure, but traditional methods itself can cause pain, making pediatric patients anxious and uncooperative in dental offices.

Effective pain management is crucial for children receiving dental injections to promote comfort, cooperation, and compliance. These techniques include topical analgesics, distraction, injection rates, buffering and warming the local anesthesia, speed reduction, fine needles, and precooling. Yet, no conclusive painless injection technique has been developed yet.

Finally, The Wand system, developed in 1997 by Milestone Scientific Inc., it was the first Computer-Controlled Local Anesthesia Delivery (CCLAD)discovered. Other devices like Morpheus, Calaject, Quicksleeper, and Smartject have entered the market, these systems varying in injection speed, design, weight, and shape, so, dentists can select the one that best meets their requirements.

This device's main concept is that a local anesthetic injection is done by lowering the pressure and flow rate.

The CCLAD reduced destructive behaviors in young children who were difficult to cooperate compared to the traditional method and created a positive experience for both the patient and physician.

The main advantage of these CCLADS devices is The ability to provide a small quantity of the local anesthetic solution with a stable injection mode, which decreases the discomfort associated with less controlled injections. In both adult and pediatric dentistry, the CCLADS devices have proven effective for extractions, pulpal therapies, and restorations. Patients also tolerate them well and behave less disruptively.

The Traditional injection syringe compared with computer-controlled local analgesic delivery devices (CCLAD) regarding disruptive behavior, pain, anxiety, and biochemical parameters. The results showed lower VAS, WBS, and salivary cortisol values in CCLADS patients compared to the traditional syringe group. They concluded that a positive impact of CCLADS on pain and anxiety can be recommended for pediatric patients.

Using CCLADs is significantly less painful than using traditional syringes and opens new, promising opportunities for working with patients presenting high dental fear.

The Starpen is one of the most recent advances that is promoted as a more comfortable and painless alternative to the traditional local anesthetic syringe. It includes a power adapter, cartridge holder, handpiece, and charging base. In dental uses, it can be injected intramuscularly or subcutaneously. It comes in three different speeds-high, low, and hybrid-and two aspiration modes-manual and auto. It may be used with the majority of the conventional gauge needles.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-8 years
* Cooperative children (Rating 3 or 4 based on the Frankl behavior scale)
* Medically fit children (ASA I).
* Children are mentally capable of communication.
* First dental visit.
* Patient requiring extraction of lower primary molars due to root caries, crown fractures, periapical disease, and failed pulpotomies.

Exclusion Criteria:

* Children with a behavioral management problem.
* Parental refusal of participation.
* Children with a previous history of local anesthesia injection.
* Medically unfit children (other than ASA I).
* Uncooperative children (other than Frankl 3,4).
* Children under medications (antibiotics and analgesics) for the previous 48 hours that could alter the pain perception.
* Teeth that showed any signs of mobility, ankylosis, or root resorption affecting more than one-third of the root

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Subjective Pain perception during injection of local anesthesia | immediately after the procedure(injection)
  After injection, the child will be asked to choose a face from the Wong-Baker faces pain rating scale to express his pain experience after explaining the scale to him (Scores from 0 to 10),The scale shows a series of faces ranging from a happy face at (0) which represents "no hurt", to a crying face at (10), which represents "hurts like the worst pain imaginable . "the higher score means a worse outcome"

SECONDARY OUTCOMES:
objective pain perception during local anesthesia injection | During the procedure (injection)
  During injection, the objective pain perception will be assisted by an external evaluator (the assistant supervisor), using the Faces, Legs, Activity, Cry, and Consolability scale with scores from (0 to 10) with score (0) represents that the patient is relaxed and comfortable and score (10) represents severe discomfort/pain "the higher score means a worse outcome"
Subjective pain perception during the extraction | immediately after the procedure(extraction)
  After extraction, the subjective pain perception will be recorded from the child by asking him to choose a face from the Wong-Baker faces pain rating scale to express his pain experience during the extraction after explaining the scale to him with scores from (0 to 10). The scale shows a series of faces ranging from a happy face at (0) which represents "no hurt", to a crying face at (10), which represents "hurts like the worst pain imaginable .
  "the higher score means a worse outcome"
objective pain perception during extraction | During the procedure (extraction)
  During extraction, the objective pain perception will be assisted by an external evaluator (the assistant supervisor), using the Faces, Legs, Activity, Cry, and Consolability scale with scores from (0 to 10) with score (0) represents that the patient is relaxed and comfortable and score (10) represents severe discomfort/pain "the higher score means a worse outcome"
Physiological parameter (heart rate) | at baseline(10 minutes before the procedure) and during both procedures (injection and extraction)
  Physiological parameter (heart rate) with measuring unit(Beats per minute ) will be recorded at three-time points: baseline (10 minutes before the procedure), during injection, and extraction with a Pulse oximeter on the child's index finger
Physiological parameter (oxygen saturation) | at baseline(10 minutes before the procedure) and during both procedures (injection and extraction)
  Physiological parameter (oxygen saturation) with measuring unit(percent (%)) will be recorded at three-time points: baseline (10 minutes before the procedure), during injection, and extraction with a Pulse oximeter on the child's index finger

REFERENCES:
- [Background] Saoji H, Nainan MT, Nanjappa N, Khairnar MR, Hishikar M, Jadhav V. Assessment of computer-controlled local anesthetic delivery system for pain control during restorative procedures: A randomized controlled trial. J Dent Res Dent Clin Dent Prospects. 2019 Fall;13(4):298-304. doi: 10.15171/joddd.2019.045. PMID 32190214
- [Background] Patini R, Staderini E, Cantiani M, Camodeca A, Guglielmi F, Gallenzi P. Dental anaesthesia for children - effects of a computer-controlled delivery system on pain and heart rate: a randomised clinical trial. Br J Oral Maxillofac Surg. 2018 Oct;56(8):744-749. doi: 10.1016/j.bjoms.2018.08.006. Epub 2018 Aug 22. PMID 30143396
- [Background] Attia S, Austermann T, May A, Mekhemar M, Conrad J, Knitschke M, Bottger S, Howaldt HP, Riad A. Pain perception following computer-controlled versus conventional dental anesthesia: randomized controlled trial. BMC Oral Health. 2022 Sep 22;22(1):425. doi: 10.1186/s12903-022-02454-1. PMID 36138388
- [Background] Janik K, Niemczyk W, Peterek R, Roj R, Balicz A, Morawiec T. Computer-Controlled Local Anaesthesia Delivery efficacy - a literature review. Saudi Dent J. 2024 Aug;36(8):1066-1071. doi: 10.1016/j.sdentj.2024.05.012. Epub 2024 May 31. PMID 39176166
- [Background] Shilpapriya M, Jayanthi M, Reddy VN, Sakthivel R, Selvaraju G, Vijayakumar P. Effectiveness of new vibration delivery system on pain associated with injection of local anesthesia in children. J Indian Soc Pedod Prev Dent. 2015 Jul-Sep;33(3):173-6. doi: 10.4103/0970-4388.160343. PMID 26156269
- [Background] Anil O, Keskin G. Comparison of computer controlled local anesthetic delivery and traditional injection regarding disruptive behaviour, pain, anxiety and biochemical parameters: a randomized controlled trial. J Clin Pediatr Dent. 2024 Jan;48(1):120-127. doi: 10.22514/jocpd.2023.046. Epub 2024 Jan 3. PMID 38239164